CLINICAL TRIAL: NCT00394576
Title: Assessing Novel Methods of Improving Patient Education of Nutrition: eHealth, Health Literacy and Chronic Kidney Disease
Brief Title: Assessing Novel Methods of Improving Patient Education of Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: H-2006-0186-1; 144-NR73 (Other Grant/Funding Number: UW Clinical Research Scholars Program); NCT00693277 (obsolete NCT alias)
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney School; Short Test of Functional Health Literacy; Chronic Kidney Disease Knowledge Assessment Tool of Nutrition; Short Form 12 version 2; Three Day Dietary Diary; Kidney Disease Self-Management Survey
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care plus Internet-based nutrition module (Experimental): usual care plus Internet-based nutrition module
  Interventions: Behavioral: Internet-based nutrition module along with usual care
- usual care (Active Comparator): usual care
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Internet-based nutrition module along with usual care — usual care plus Internet-based nutrition module
  Arms: usual care plus Internet-based nutrition module
Behavioral: usual care — usual care
  Arms: usual care

SUMMARY:
The relationship between elevated phosphorus levels and morbidity and mortality in patients with chronic kidney disease (CKD) is well recognized, and dietary phosphorus restriction is a mainstay of phosphate management. Current study is an effort to test the effect of a web-based nutritional educational intervention, Kidney School(KS), to improve phosphorous knowledge and control phosphorous intake in CKD patients.

DETAILED DESCRIPTION:
The relationship between elevated phosphorous level in the severity of Chronic kidney disease(CKD) is well documented. However, appropriate control of phosphate intake remains sub-par, due in part to the difficulties that patients have understanding phosphate content in foods.

Randomized trials have shown that intensive, individualized dietary counseling can improve patient knowledge about phosphorus and help control hyperphosphatemia; however, maintaining this level of counseling is time-consuming, costly, and impractical. Given the recognized nephrology workforce shortage, there is a crucial need for systems to fill this gap with novel technologies to educate patients, and it is vital that a better understanding of the effects of novel nutritional intervention counseling methods on patient knowledge, nutritional intake and nutritional status be evaluated in CKD patients.

Furthermore, to effectively engage in the patient side of the education process, those who receive it, the patients, must be able to comprehend information and draw on it for decision-making. Novel educational interventions may be better suited than traditional methods to circumvent literacy limitations. Therefore, it is vital to assess the relation of functional health literacy of this population in both traditional and emerging educational venues.

Kidney School (KS, http://www.kidneyschool.org) is an online, personalized, interactive self-management learning center created by the Madison, WI based Medical Education Institute (MEI) and organized into fifteen 20-30 minute modules, each focused on a different topic related to kidney disease and its treatment, including nutrition. Content is based on 10 years of research conducted by the Life Options Rehabilitation Program, with internal and external expert review. The nutrition module is tailored for patients with or without diabetes.

The importance of phosphorus control for patients with CKD has traditionally been vital to prevent bone disease. More recently it is recognized that poor phosphorus control correlates with cardiovascular disease, of which patients with CKD carry an enormous burden. Similarly, there has recently been much attention to circulating endothelial cells (CECs) as a novel marker for cardiovascular risk in this population. While the ultimate test would be to determine if controlling phosphorus impacts on cardiovascular events, that is beyond the scope of this project. Therefore, we propose to measure levels of CECs as an intermediary step toward cardiovascular events, in correlation to phosphorus intake.

Following enrollment and informed consent, subjects will be randomized to one of two arms [group1: usual care; group 2: usual care plus Kidney School (KS)].

Kidney School (KS, http://www.kidneyschool.org) is an online, personalized, interactive self-management learning center created by the Madison, WI based Medical Education Institute (MEI) and organized into fifteen 20-30 minute modules, each focused on a different topic related to kidney disease and its treatment, including nutrition. Content is based on 10 years of research conducted by the Life Options Rehabilitation Program, with internal and external expert review. The nutrition module is tailored for patients with or without diabetes.

Proprietary Information. The mission of the non-profit MEI is to help people with chronic diseases learn to manage and improve their health, through research and education. The MEI believes charging a fee for educational materials can be a barrier between patients and the information they need to live successfully with a chronic disease. All MEI-developed patient education materials are therefore free. KS is entirely proprietary to the MEI, but will continue to be available free of charge via the Internet. KS is fully compliant with HIPAA standards.

The SF-12 Health Survey version 2 is a 12-item measure of health related quality of life. Widely used in research in a variety of disease states, including CKD, it provides physical and mental component summary scores with a strong concordance with the lengthier SF-36. Given that we will be administering multiple cognitive and behavioral surveys to subjects, the shorter version will be used.

Kidney Disease Self-Management Survey (KDSMS). Developed by MEI, the KDSMS is a 58-item Likert scale with 6 subscales, based on theories deemed important for self-management education in other chronic diseases, including the health belief model, self-efficacy, behavioral intent, and the transtheoretical model. These theories converge into a self-management education schema that emphasizes the importance of information, support, modeling, planning, practice and monitoring, and reflection in patient self-management education. The 6 subscales are: 1) Self-monitoring, 2) Adjusting to symptoms, 3) Lifestyle behaviors, 4) Medication-taking, 5) Information seeking, 6) Doctor/patient communication.

24 hour recall diaries - After collecting the information from subjects, nutrient analysis will be performed using The Food Processor SQL Nutrition Software (ESHA Research, Salem, Oregon).

The study instruments will all performed for research purposes. While some of them (the S-TOFHLA, 3-Day Dietary Diaries) have been used as part of patient care, this is not routine, and it is not done at our facilities.

Lab work collected will consist of serum phosphorus, calcium and intact-parathyroid hormone levels. As these are routinely collected prior to or during a regular CKD clinic visit, the study coordinator will check to see if this data is already available, and will not duplicate this blood work if it is. In addition, all subjects will have blood drawn (30 ml) for assessment of circulating endothelial cells (CECs), a novel marker for vascular damage.

Following baseline data collection, group 1 will continue with their scheduled clinic visit, while group 2 will spend approximately 30 minutes completing the KS nutrition module at a dedicated computer education station at the UW Kidney Clinic. The study coordinator will bring up the KS nutrition module (tailored for diabetes as a co-morbidity if appropriate). After completion of the KS nutrition module, patients will receive a personalize action plan, and then proceed with their scheduled clinic visit.

All subjects will then be asked to return in 30-60 days to repeat some of the survey information and blood work.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 and less than 90
* Chronic kidney disease stage 3, 4 or 5
* Adequate visual acuity with correction to allow discrimination of 14-point type
* Ability to read English
* Ability to provide informed consent

Exclusion Criteria:

* Anticipated need for renal replacement therapy within 60 days
* Prison population

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Gain in phosphorus knowledge as assessed by the chronic kidney disease Knowledge Assessment Tool (CKDKAT) of nutrition. | 4 to 8 weeks post intial questionnaire/survey
  The CKDKAT of nutrition is a revised version of the original CKDKAT, which addresses only nutritional knowledge specific to chronic kidney disease (CKD). 15 of 25 questions are phosphorus-specific, with the remaining 10 concerning sodium, potassium and protein intake.
Compliance with dietary phosphorous will be measured by serum phosphorous level. | 4 to 8 weeks after initial questionnaire/survey appointment
  Measurement of compliance with dietary phosphorous will be measured by serum phosphorous level. In CKD, Phosphorus excretion diminishes, leading to an increase in serum phosphorus levels.
Compliance with dietary phosphorous will be measured by serum calcium level | 4 to 8 weeks after initial questionaire/survey appointment
  Measurement of compliance with dietary phosphorous will be measured by serum calcium level. In CKD, calcium is not reabsorbed, leading to decreased serum calcium.
Compliance with dietary phosphorous will be measured by para thyroid hormone (PTH) level | 4 to 8 weeks after initial questionnaire/survey appointment
  Measurement of compliance with dietary phosphorous will be measured by para thyroid hormone (PTH) level. In CKD, Both decreased serum calcium levels and increased serum phosphorus levels stimulate excessive secretion of PTH.
Compliance with dietary phosphorous will be measured by serum calcium phosphorus product. | 4 to 8 weeks after initial questionnaire/survey appointment
  Measurement of compliance with dietary phosphorous will be measured by serum calcium phosphorus product.
Compliance with dietary phosphorus intake will be measured by using 24 hour recall diary. | 4 to 8 weeks after initial questionnaire/survey appointment
  For measuring compliance with dietary phosphorus intake, data will be collected by 24 hour recall diaries. Nutrient analysis data will be analyzed by Food Processor SQL Nutrition Software (ESHA Research, Salem, Oregon)

SECONDARY OUTCOMES:
Correlations between dietary phosphorus intake, serum phosphorous levels and circulating endothelial cells (CECs) in CKD | 2 years
  After all groups have completed their visits, correlations between dietary phosphorus intake, serum phosphorous levels and CECs will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Jaffery, MD, Principal Investigator — School of Medicine and Public Health, University of Wisconsin
Locations (1):
- UW Health Kidney Clinic and Wisconsin Dialysis, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- See also: Kidney School(KS) is an online, personalized, interactive self-management learning center created by the Madison, WI based Medical Education Institute (MEI) — http://www.kidneyschool.org